CLINICAL TRIAL: NCT02785614
Title: Pharmacokinetics Study of Trazodone Hydrochloride Prolonged-Released Tablets in Chinese Healthy Volunteers
Brief Title: PK Study of Multi-dose Trazodone Hydrochloride Prolonged-released Tablets in Healthy Chinese
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Zhaoke-201603-Tra-Trial II
Record Dates: First submitted 2016-05-24; First posted 2016-05-30 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Trazodone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- II-1 (Experimental): This is 2-period, 2 cross (2x2) crossover design was used. each 3 males and 3 females, give the following two different crossover treatments in the following sequence:
  R: trazodone hydrochloride tablets 50mg for 3 times per day for 7 days T: trazodone hydrochloride prolonged-release tablets 150 mg per day for 7 days. Wash-out period is 14 days.
  Interventions: Drug: trazodone hydrochloride prolonged-release tablet; Drug: trazodone hydrochloride tablet
- II-2 (Experimental): This is 2-period, 2 cross (2x2) crossover design was used. each 3 males and 3 females, give the following two different crossover treatments in the following sequence:
  T: trazodone hydrochloride prolonged-release tablets 150 mg per day for 7 days R: trazodone hydrochloride tablets 50mg for 3 times per day for 7 days. Wash-out period is 14 days.
  Interventions: Drug: trazodone hydrochloride prolonged-release tablet; Drug: trazodone hydrochloride tablet

INTERVENTIONS:
Drug: trazodone hydrochloride prolonged-release tablet — 150 mg, oral administration, 1 per day
Drug: trazodone hydrochloride tablet — 50mg, oral administration 3 times per day

SUMMARY:
The main objective is to evaluate the pharmacokinetics comparative studies in a single dose, multiple dose

DETAILED DESCRIPTION:
Trial II Multiple dose, the highest specification (150mg) pharmacokinetic study of Trazodone Hydrochloride Prolonged Release Tablets; 12 patients (males and females, half and half).

2-period, 2 cross (2x2) crossover design was used. screened 12 subjects (males and females) were randomly divided into two groups (II-1、II-2), each 3 males and 3 females, give the following two different crossover treatments: trazodone hydrochloride prolonged-release tablets 150 mg per day for 7 days in T group, trazodone hydrochloride tablets 50mg for 3 times per day for 7 days in R group. Wash-out period is 14 days.

Trial II. 2X2 design Group Period 1 Period 2 II -1 R T II -2 T R T group: the subjects will be provided trazodone hydrochloride prolonged-release tablet 150mg at about8:00am each day. Sampling site will be conducted in day 1, 5, 6, 7 before administration in this period, blood sampling will be conducted in 0.5, 1.0, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36.0, 48.0, 72.0h after administration on day 7.

R group: The subjects will receive 50mg trazodone hydrochloride tablet 50mg for 3 times after receiving standard light breakfast at 6:00am, standard meal at 14:00 and 22:00. Blood sampling will be conducted on day 1, 5, 6, 7 before first administration in this period, blood sampling will be conducted at 0.5, 1.0, 1.5, 2.0, 3.0, 4.0, 6.0, 8.0 (before the second time administration), 8.5, 9.0, 9.5, 10.0, 11.0, 12.0, 14.0, 16.0 (before the third time administration), 16.5, 17.0, 17.5, 18.0, 19.0, 20.0, 22.0, 24.0, 36.0, 48.0, 72.0h after administration on day 7.

5.0 mL venous blood from forearm venous blood was took through venous indwelling needle and transfer into the heparin tube. After plasma separation it stored in low temperature in a refrigerator.

ELIGIBILITY:
Inclusion Criteria:

* Weight: all the subjects should be≥50 kg, BMI within 19~24 kg/m2
* Blood pressure: SBP 90-140mmHg，DBP 50-90 mmHg；
* All the subjects should understand this trial well and sign the inform consent form before participating this study;
* Subjects should be able to communicate with investigators well and complete this study in accordance with protocol.

Exclusion Criteria:

* The baseline value of safety evaluation index is considered to be abnormal with clinical significance by investigators before participating the trial.
* A positive hepatitis B surface antigen result；
* A positive hepatitis C surface antigen result；
* A positive test for HIV antibody and syphilis testing；

Any of the abnormalities of ECGs examination occurs in screening period or the first day of administration:

* With the history of using any drug which will inhibit or induce liver to metabolize drug within 1 month before the study initiation;
* With the history of administrating any drugs (prescription medicine, over-the-counter drug and Chinese herbal medicine) within 2 week before the study initiation;
* Past history of heart disease, cardiac failure, myocardial infarction, angina, unknown cause of arrhythmia, point swinging pattern of ventricular tachycardia, ventricular tachycardia, long QT syndrome or long QT syndrome and family history (with genetic proof or there were any close relatives died because of heart disease);
* History of thyroid disease or past history of thyroid surgery;
* History of immune system disease (such as thymus disease)；
* With surgery history within 6 months before this study initiation；
* History of severe digestive disease (such as gallbladder disease with significant clinical significance, jaundice or susceptive jaundice, hepatocellular adenoma, hepatic cavernous hemangioma and the other liver diseases)；
* With history of gastrointestinal, liver and renal disease (no matter it has been cured or not) which will affect drug absorption and metabolism within 6 months before this study initiating
* History of any serve cardiocerebral vascular system, respiratory system, metabolic system and nervous system diseases;
* History of hematological system diseases, such as coagulation disorders；
* History of tumor；
* Subjects with hypokalemia and hypocalcemia (according to the lower limit value of the laboratory reference ranges；

Life style:

* History of alcohol addicted within 6 months before the study
* Smoking >1 cigarettes a day in the last 3 months prior to this study;
* History of drug abuse and taking drugs (such as marihuana, cocaine, opium, benzodizepines, amphetamines, barbiturates, tricyclic antidepressant).
* History of consumption of excessive tea, coffee and/or caffeinated beverage (more than 8 cups/day) within the period of 2 days before the administration and 8 days after administration.
* History of consumption of grapefruit juice within the period of 2 days before and 8 days after administration.

Others：

* Subjects who reject to take effective contraceptive measures within the time period after inclusion to 3 months after administration;
* Subjects with allergic constitution, including those who are allergic to the excipient (microcrystalline cellulose, lactose, aerosil, sodium carboxymethyl starch, magnesium stearate) of this product;
* History of participating any clinical trial within 3 months before this study, or participating the other clinical trial within the time period of inclusion to one month after the last time visit(after the last time administration);
* History of blood donation within 3 months prior to this study, or within the time period of inclusion to one month after the last time visit (after the last time administration);
* Subjects who have food allergy or have any special diet requirements, or who cannot follow the standard diet;
* Subjects who, in the opinion of the investigator, should not participate in the study；

The female subjects are not eligible for inclusion in this study if she meet any of the following criteria above and below:

* With the history of consumption of oral contraceptive within one month prior to this study；
* History of long-acting estrogen or progesterone injection or implant within 6 months prior to this study;
* The bearing-age female subjects who have not taken appropriate contraceptives within 2 weeks prior to this study;
* The bearing-age female subjects and their spouse are not willing to take the following contraceptives measure, condom, copper intrauterine device within 3 months after inclusion;
* Subjects who are in gestation period and lactation period;
* Subjects with positive hCG test;
* Single menstrual more than 80ml.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-01-04 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | day 1, 5, 6, 7 before administration and 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 16 hours, 20 hours, 24 hours, 36 hours, 48 hours, 72 hours after administration on day 7
  To observe area under curve characteristics of Trazodone in single or multiple dose groups

CONTACTS AND LOCATIONS:
Locations (1):
- Phase I Clinical Trial Centre, Chinese University of Hong Kong, Hong Kong, Sha Tin New Territories, Hong Kong